CLINICAL TRIAL: NCT00870909
Title: Anodal & Cathodal tDCS for Treatment of Resistant Auditory Hallucinations in Schizophrenia
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-A01226-49
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia; Auditory Hallucinations
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS (Active Comparator): tDCS active; - Intensity = 2 milliamps (mA) during 20 minutes. ramp up/ramp down 30sec anodal tDCS applied over the left DLPFC combined with cathodal tDCS applied over the left temporoparietal junction (TPJ).
  10 sessions, 2 per day
  Interventions: Procedure: active tDCS
- sham tDCS (Placebo Comparator): tDCS placebo same electrode montage than in the active group. 30 sec of active tDCS in the beginning of the stimulation sessions; ramp up/ramp down 30 sec
  Interventions: Procedure: sham tDCS

INTERVENTIONS:
Procedure: active tDCS — Intensity 2 mA during 20 minutes, 2 times per day
  Other Names: tDCS; transDirect Current Stimulation; Anodal tDCS; Cathodal tDCS
  Arms: active tDCS
Procedure: sham tDCS — sham condition as delivered by the stimulator
  Other Names: tDCS placebo
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to determine whether trans Direct Current Stimulation (tDCS) is effective in the treatment of auditory hallucinations in schizophrenia.

DETAILED DESCRIPTION:
The project will investigate the use of a novel technique, transcranial direct current stimulation (tDCS) in the treatment of patients with schizophrenia. tDCS permit the application of an extremely weak continuous electrical current to the brain through an anode and a cathode applied on the scalp. Anodal stimulation appears to increase brain activity whereas cathodal stimulation has the opposite effect.

Using anodal & cathodal tDCS the investigators aimed to treat auditory hallucinations, a symptoms of schizophrenia. The investigators plan to apply tDCS such that it can simultaneously increased activity in the frontal brain areas and reduce activity over temporoparietal cortex, 2 areas involved in the physiopathology of the disease. Real active stimulation will be compare to a sham condition in 60 patients (30 in each group). 30 patients will be included in a French center (Hospital le Vinatier, sponsor of the study) and 30 in Tunisia (laboratory "vulnerability to psychosis" (Pr Gaha) à Monastir).

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia according to Diagnostic and Statistical Manual - DSM-IV
* Auditory verbal hallucinations for at least 6 weeks (despite antipsychotic drugs)
* Medication Resistance according to Kane et al., 1988
* Age between 18 and 50 years old
* Informed consent

Exclusion Criteria:

* Concomitant major and unstable medical or neurologic illness
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2016-04-21 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Auditory hallucinations measured by Auditory Hallucination Rating Scale (Hoffman et al., 2003) | before, after 1 week of treatment and 2 times follow up (1 & 3 months)

SECONDARY OUTCOMES:
Neurochemical impact of treatment measured by 1H-MRS (proton Magnetic Resonance Spectroscopy), DTI (Diffusion Tensor Imaging) and resting MRI | 3 times: before treatment, immediately after treatment and a last evaluation 1 month after

CONTACTS AND LOCATIONS:
Overall Officials: emmanuel poulet, MD, PhD, Principal Investigator — Hopital Le Vinatier; JEROME BRUNELIN, PhD, Study Director — Hopital le Vinatier
Locations (2):
- Hopital Le vinatier, Bron, France
- Laboratoire de Recherche " Vulnérabilité Aux Psychoses ", Monastir, Tunisia

REFERENCES:
- [Derived] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236